CLINICAL TRIAL: NCT02531425
Title: Evaluation of Pharmacodynamic Effects of Intratumoral Delivery of Plasmid IL-12 Electroporation in Patients With Triple Negative Breast Cancer
Brief Title: Evaluation of Pharmacodynamic Effects of IT-pIL12-EP in Patients With TNBC
Acronym: TNBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I140
Record Dates: First submitted 2015-08-18; First posted 2015-08-24 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: ER-Negative PR-Negative HER2-Negative Breast Cancer
Keywords: TNBC; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IT-pIL12-EP (Experimental): intratumoral injection of plasmid-IL12 following immediately by electroporation
  Interventions: Biological: IT-pIL12-EP

INTERVENTIONS:
Biological: IT-pIL12-EP — Intratumoral pIL-12 injections followed immediately by electroporation into accessible tumor lesions
  Other Names: intratumoral plasmid-IL-12 + Electroporation

SUMMARY:
Intratumoral plasmid IL-12 electroporation (IT-pIL12-EP) will be administered to approximately 10 patients with triple negative breast cancer (TNBC) with cutaneous or subcutaneous disease. Patients will receive one complete cycle of therapy, consisting of local injection of plasmid IL-12 (pIL-12) followed immediately by electroporation (EP), into accessible tumor lesions. IT-pIL12-EP will be administered in Days 1, 5, and 8 of the single 28-day cycle.

DETAILED DESCRIPTION:
This pilot study will evaluate the pharmacodynamic effects of intratumoral injection of pIL-12 followed immediately by electroporation (IT-pIL12-EP). A minimum of ten patients with biopsy-accessible triple negative breast cancer (TNBC) will be treated in this study. Additional patients, up to a maximum of 25 patients, may be enrolled based upon pharmacodynamic observations and at the discretion of the Principal Investigator, in consultation with the Sponsor. All patients will receive a single 28-day treatment cycle. One lesion will remain untreated (the control lesion). Treatment will be administered on Days 1,5, and 8 of the single 28-day cycle. Treatments will consist of direct injection of pIL-12 into tumor lesions, followed immediately by electroporation of the lesions. At the end of the treatment cycle, patients will return to clinic for a final safety evaluation and tumor biopsy. This end of study (EOS) visit will occur prior to initiating any new anti-cancer therapy/regimen.

All patients will undergo tumor biopsies at two separate timepoints for molecular and histological analyses associated with the primary endpoint. At least one lesion will be biopsied at Screening (pre-treatment sample). Biopsies of the untreated control lesion and at least one treated lesion will be obtained at the EOS visit (post-treatment samples). Additional tumor biopsy samples may be requested if there is either tumor regression or progression prior to EOS.

Duration of participation will be approximately 4 weeks for each patient. A patient is considered to have completed the study if all three IT-pIL12-EP treatments (Days 1, 5, & 8) and all required pre- and post-treatment tumor biopsies have been obtained and EOS safety follow-up evaluations have been performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of locally-advanced, inoperable, metastatic and/or treatment-refractory triple negative breast cancer (TNBC). *Treatment refractory disease is defined as the persistence of tumor lesions following at least one intervention that may include chemotherapy, radiation and/or surgery, or any combination thereof. *Patients must have both ER and PR staining < 5% and be HER2-negative. Patients with ER or PR staining of 5-10%, but who have historically been treated as TNBC may also be enrolled. *Patients must not have disease that, in the opinion of the investigator, is considered amenable to potentially curative treatment.
* Age ≥ 18 years.
* ECOG Performance Status of 0-1.
* Life expectancy ≥ 6 months.
* Patients may have had radiation therapy, but must have progressive disease after radiation therapy if the lesions to be treated are within the radiation field. Radiation treatment must be completed ≥ 4 weeks prior to Cycle 1 Day 1.
* Adequate hepatic function with total bilirubin and ALT < 1.5X the upper limit of normal (ULN), except in patients with Gilbert's Syndrome must have a total bilirubin < 3X ULN and ALT < 3X ULN. In cases of known liver metastases, ALT ≤ 5X ULN is acceptable (total bilirubin must be < 1.5X ULN).
* Adequate renal function, estimated or calculated creatinine clearance of > 50 mL/min (calculated using the formula of Cockcroft and Gault) -or- serum creatinine ≤ 2.0 mg/dL.
* Adequate hematological function, defined as ANC ≥ 1,500/mm3, Hb ≥ 9.0 g/dL, and platelet count ≥ 100,000/mm3.
* Lesions that are accessible for injection and electroporation, defined as cutaneous or subcutaneous disease.
* At least 2 anatomically distinct lesions accessible for biopsy.
* Must consent to study-specific biopsies at two separate timepoints: pre-treatment (Screening) and post-treatment (Day 28 or EOS).
* Tumor lesions in the CNS are permitted but lesions must have been stable for at least 3 months prior to Cycle 1 Day 1 (C1D1). Stable CNS lesions are defined as not requiring steroid prophylaxis or other medications to prevent seizures or other complications associated with CNS lesions and no evidence of worsening of CNS disease.
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to C1D1 and agree to use dual methods of contraception during the study and for a minimum of 30 days following the last treatment. Post menopausal females (>45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements.

Male patients must use an effective barrier method of contraception during the study and for a minimum of 30 days following the last treatment if sexually active with a female of childbearing potential.

* Resolution of all treatment-related toxicities, except alopecia, anemia and neuropathy, from any previous cancer therapy to ≤ Grade 1 prior to the first dose of study treatment.
* Ability to provide written informed consent.

Exclusion Criteria:

* Any other current or previous malignancy within the past three years that, in the opinion of the Principal Investigator, will interfere with study-specific objectives.
* Patients with electronic pacemakers or defibrillators.
* Chemotherapy or hormonal therapy for anti-cancer treatment within 28 days prior to Cycle 1 Day 1.
* Immunotherapy or biological therapy (e.g., monoclonal antibodies) within 28 days prior to Cycle 1 Day 1, unless pre-approval is obtained from the Sponsor Medical Monitor.
* Treatment with unapproved investigational therapeutic agent within 28 days prior to Cycle 1 Day 1, unless pre-approval is obtained from the Sponsor Medical Monitor.
* Patients receiving systemic steroid therapy for a chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's Disease, etc.). Topical steroids are also excluded. Nasal and inhaled steroids are permitted.
* Unstable/inadequate cardiac function:

  * symptomatic ischemia
  * uncontrolled or clinically significant conduction abnormalities; first degree AV block or asymptomatic LAFB/RBBB are eligible
  * myocardial infarction in the previous six months
  * congestive heart failure (New York Heart Association class III to IV)
* Major surgery within 28 days prior to C1D1.
* Infection requiring parenteral antibiotics, antivirals, or antifungals within 2 weeks prior to C1D1.
* Patients who are known to have HIV infection/seropositivity.
* Active Hepatitis A, B, or C infection or known to be positive for HCV RNA or HBV surface antigen. Patients who have been vaccinated against Hepatitis B and who are positive for ONLY the Hepatitis B surface antibody are permitted to participate in the study.
* Serious psychiatric or medical conditions that could interfere with treatment or protocol-related procedures.
* Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in the proportion of intratumoral lymphocyte subsets | 28 days
  Paired tumor biopsy samples will be quantitatively analyzed for the number and distribution of tumor infiltrating lymphocytes (TILs).
NanoString-based gene expression | 28 days
  Comparison of NanoString-based gene expression profiles will be completed from paired tumor samples obtained pre- and post-treatment

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as assessed by the CTCAE v4.0 | 28 days
  Patients will be evaluated throughout study participation with physical exams and standard clinical laboratory tests (e.g., hematology, serum chemistry) for the occurrence of adverse events. The incidence and severity of treatment-related adverse events will reported using descriptive statistics.
Anti-tumor activity | 28 days
  Describe evidence of anti-tumor activity
Detection of plasmid IL-12 in untreated lesions | 28 days
  Assessment of plasmid IL-12 expression for biodistribution evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Sharron Gargosky, PhD, Study Director — OncoSec Medical Incorporated
Locations (1):
- Stanford University, Stanford, California, United States